CLINICAL TRIAL: NCT06028022
Title: Reishi Mushroom Extract for Fatigue and/or Arthralgias in Patients With Breast Cancer on Aromatase Inhibitors: A Randomized Phase II MNCCTN Trial
Brief Title: Reishi Mushroom Extract for Fatigue and/or Arthralgias/Myalgias in Patients With Breast Cancer on Aromatase Inhibitors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: MC221002; NCI-2023-06578 (Registry Identifier: CTRP (Clinical Trials Reporting Program)); MC221002 (Other: Mayo Clinic in Rochester); 23-005266 (Other: Mayo Clinic Institutional Review Board); MNCCTN032 (Other: Minnesota Cancer Clinical Trials Network)
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Estrogen Receptor-Positive Breast Carcinoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Reishi mushroom extract, placebo) (Experimental): Patients receive Reishi mushroom extract PO TID on days 1-28 for weeks 1-4 and then placebo PO TID on days 1-28 for weeks 5-8 in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: Mushroom Extract; Drug: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (placebo, Reishi mushroom extract) (Experimental): Patients receive placebo PO TID on days 1-28 for weeks 1-4 and Reishi mushroom extract PO TID on days 1-28 for weeks 5-8 in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: Mushroom Extract; Drug: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Dietary Supplement: Mushroom Extract — Given Reishi mushroom extract PO
  Other Names: Agaricus bisporus Extract; Cultivated Mushroom
Drug: Placebo Administration — Given PO
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests how well Reishi mushroom extract works in treating fatigue and/or joint/muscle pain (arthralgias/myalgias) in patients with breast cancer on aromatase inhibitors. Fatigue and arthralgias/myalgias are common symptoms in breast cancer patients taking aromatase inhibitors (AI). Given the long duration of AI treatment for some women (up to 10 years), these symptoms can significantly impact quality of life and premature discontinuation of AIs, a beneficial medication. Reishi mushrooms are among several medicinal mushrooms that have been used for hundreds of years, mainly in Asian countries, to help enhance the immune system, reduce stress, improve sleep, and lessen fatigue. Reishi mushroom extracts have not been studied explicitly for treatment-induced arthralgias/myalgias, but have been shown to improve quality of life, muscular strength, pain, and flexibility. Information from this study may help researchers determine the effect of Reishi mushroom extract on fatigue and arthralgias/myalgias in breast cancer patients receiving an AI.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of 1,000 mg three times daily (TID) of Reishi mushroom extracts as therapy for cancer-related fatigue measured by uniscale measurement at the end of four weeks.

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of Reishi mushroom extracts as therapy for cancer-related arthralgias at the end of four weeks and four weeks after cross-over as measured by the Brief Pain index (BPI)-adapted for AI associated arthralgias.

II. To evaluate the effect of Reishi mushroom extracts on cancer-related quality of life (QOL), as measured by uniscale, at the end of four weeks and four weeks after cross-over.

III. To evaluate the efficacy of Reishi mushroom extracts on mood, as assessed by the World Health Organization Five Well-Being Index (WHO-5) item well-being scale, at the end of four weeks and four weeks after cross-over.

IV. To evaluate treatment toxicity between the two treatment arms, as measured by a patient symptom experience diary and weekly calls from the study team.

V. To evaluate the interest, knowledge, and acceptance of integrative treatments for cancer-related symptoms.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive Reishi mushroom extract orally (PO) TID on days 1-28 for weeks 1-4 and then placebo PO TID on days 1-28 for weeks 5-8 in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo PO TID on days 1-28 for weeks 1-4 and Reishi mushroom extract PO TID on days 1-28 for weeks 5-8 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* History of breast cancer, estrogen receptor positive (ER+), Her 2 positive or negative
* Fatigue ≥ 4/10
* Currently post-menopausal (as defined by National Comprehensive Cancer Network (version 4.2024), taking any aromatase inhibitor in the curative setting and planning to be on such for at least 8 weeks after registration. [Patients on concurrent ovarian suppression (such as with leuprolide acetate, goserelin) are allowed]; CDK 4/6 inhibitors abemaciclib, ribociclib ARE allowed
* Prior treatment: last chemotherapy ≥ 90 days prior to randomization (if treated with chemotherapy)
* On a stable dose of pain medications if pain medications are being regularly used. (i.e., no change in dosage in the past 30 days)
* If on supplements, must be on stable dose with no plan to change; not on or planning any acupuncture or other specific supportive modalities for fatigue or AI arthralgias
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* White blood cell count (WBC) ≥ 3,000/mm^3 (obtained ≤ 30 days prior to randomization)
* Hemoglobin ≥ 10 g/dL (obtained ≤ 30 days prior to randomization)
* Platelet count ≥ 100,000/mm^3 (obtained ≤ 30 days prior to randomization)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (obtained ≤ 30 days prior to randomization)
* Alanine aminotransferase (ALT) or aspartate transaminase (AST) ≤ 1.2 x ULN (obtained ≤ 30 days prior to randomization)
* Prothrombin time (PT)/activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN (obtained ≤ 30 days prior to randomization)
* Negative pregnancy test done ≤ 7 days prior to registration, for persons on concurrent ovarian suppression only
* Provide informed consent
* Ability to complete questionnaires
* Willing to return to enrolling institution during the active monitoring phase of the study
* Patients who have had a recent surgery or procedure should be healed and cleared by their clinician and/or surgeon per local standards, prior to registration

Exclusion Criteria:

* Other known uncontrolled medical conditions causing fatigue such as untreated thyroid disease, depression, fibromyalgia, chronic fatigue syndrome, infection, autoimmune disease, or active/untreated hepatitis
* Allergy to mushrooms
* On anticoagulation medication or aspirin or having a known bleeding disorder
* On any specific medication for fatigue (e.g., methylphenidate)
* Metastatic cancer diagnosis (history of nodal metastases is allowed)
* Chronic steroid use, unless on physiologic replacement doses
* Current use of any medical mushrooms
* On medications for diabetes
* History of symptomatic hypotension
* Taking CYP3A4, CYP2D6 sensitive substrates which can be located at the following link:

https://www.fda.gov/drugs/drug-interactions-labeling/healthcare-professionals-fdas-examples-drugs-interact-cyp-enzymes-and-transporter-systems

* Drugs which exhibit either >20% inhibition or >20% induction of CYP2E1 in vivo, such as: Acetaminophen, Dapsone, Enflurane, Halothane, Isoflurane, & Theophylline
* Taking olaparib
* Any of the following because this study involves an agent that has unknown genotoxic, mutagenic and teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Persons on concurrent ovarian suppression who are unwilling to employ adequate contraception (e.g., hormonal methods, barrier methods, intrauterine device, abstinence)
* Planned surgery or procedure during time on study and ≤ 14 days after last dose, due to bleeding risks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2026-10-16 (Estimated); Study Completion 2026-10-16 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue scores | Baseline to end of four weeks
  Based on a single item fatigue uniscale question. Will be compared between arms using a two-sided two-sample t-test assuming equal variances in each group.

SECONDARY OUTCOMES:
Change in quality of life | Baseline to the end of four weeks and four weeks after cross-over
  Measured by the World Health Organization-Five Well-Being Index. Will be compared between arms using two-sample, two-sided t-tests assuming equal variances and alpha levels of 5%. The analyses of the crossover portion of the study will be descriptive. Mean values will be plotted over time by arm. A formal crossover analysis will also be performed using Senn's linear modeling approach.
Change in arthralgias | Baseline to the end of four weeks and four weeks after cross-over
  Measured by the Brief Pain Inventory for Aromatase Inhibitor Induced Arthralgia. Will be compared between arms using two-sample, two-sided t-tests assuming equal variances and alpha levels of 5%. The analyses of the crossover portion of the study will be descriptive. Mean values will be plotted over time by arm. A formal crossover analysis will also be performed using Senn's linear modeling approach.
Incidence of adverse events | Up to 30 days follow-up
  Measured by the symptom experience diary. Will be compared between arms using two-sample, two-sided t-tests assuming equal variances and alpha levels of 5%. The analyses of the crossover portion of the study will be descriptive. Mean values will be plotted over time by arm. A formal crossover analysis will also be performed using Senn's linear modeling approach.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy D. D'Andre, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (23):
- United States (23):
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Essentia Health Baxter Clinic, Baxter, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Ely Clinic, Ely, Minnesota
  - Essentia Health Fosston, Fosston, Minnesota
  - Fairview Grand Itasca Clinic & Hospital, Grand Rapids, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Range Medical Center, Hibbing, Minnesota
  - Essentia Health International Falls Clinic, International Falls, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - MMCORC CentraCare Monticello Cancer Center, Monticello, Minnesota
  - Essentia Health Moose Lake, Moose Lake, Minnesota
  - Essentia Health Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Sanford Worthington Medical Center, Worthington, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials